CLINICAL TRIAL: NCT04603235
Title: Manual-based Art Therapy for Adolescents With Depression: a Pilot Study in Child and Youth Psychiatric Clinic in Sweden
Brief Title: Manual-based Art Therapy for Adolescents With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Child and Adolescent Psychiatry, Stockholm (Industry)
Responsible Party: Principal Investigator, Christina Blomdahl, Research and Development manager, Vastra Gotaland Region
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 254011
Record Dates: First submitted 2020-06-29; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Depression; Depressive Disorder
Keywords: art therapy; program development; Adolescent Health
MeSH Terms: conditions — Depression; Depressive Disorder

STUDY DESIGN:
Masking Description: The participants identities are masked for researchers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): This is a quasi-experimental study
  Interventions: Behavioral: Manual-based Art Therapy

INTERVENTIONS:
Behavioral: Manual-based Art Therapy — This is a manual-based treatment and consists of 10 one-hour weekly sessions. The treatment consist of detailed guidelines based on phenomenological art therapy. The sessions follow the same structure: Introduction, short relaxation, art-making, reflections about the image, and conclusions. Examples of comprised art tasks; lifeline, emotional scribbles, and different roles. The art tasks served as a prompt for painting.

SUMMARY:
There is a need to evaluate different interventions in order to meet young people's needs of treatment. The study's goal is to find out if manual-based art therapy is a useful method for young people with depression and thus increase the availability of methods of treatment for adolescents with depression in Child and youth psychiatry in Sweden.

The aim is to investigate whether manual-based art therapy is useful as treatment for adolescents with depression by examining feasibility, acceptability and compliant to treatment. Secondary, preliminary study of adolescent depressive symptoms, quality of life and functional level is affected by the treatment.

Method: Data from youths aged 13-17 years old and their parents will be collected with questionnaires and structured interviews. Measurements are taken before and after treatment. Acceptability and feasibility will be examined by participants' presence, drop out and cancellations and also by checking the art therapists' compliance to the manual and investigate their reasons to diverge from the manual

ELIGIBILITY:
Inclusion Criteria:

* Age 13-17 year
* Depression as main diagnosis

Exclusion Criteria:

* high suicide risk
* ongoing psychosis
* eating disorder
* Untreated PTSD
* Patients are excluded if there is suspicion of violence, abuse, abuse in the home or other vulnerability which requires other interventions to ensure the safety.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
Adherence to manual - therapists | 10 weeks
  the therapists self-rate their compliance to the manual on a 4 point Likert scale. describing reasons to adverting from manual
Change of Treatment satisfaction | Change from baseline at 10 weeks
  Level of satisfactions rated on a 5 point Likert scale. Higher scores indicates higher satisfaction.

SECONDARY OUTCOMES:
Change of Depression with Beck Depression Inventory BDI-II | Change from baseline at 10 weeks
  contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher score indicate more severe depression.
Change of quality of life measured with KIDSCREEN-10 | Change from baseline at 10 weeks
  Measure global Health related quality of life. HRQoL score for monitoring and screening uses. the questionnaire consist of 10 questions, each answer being scored on a 5 points Likert scale.
Change of functional impairment measured with Education,Work and Social adjustment Scale EWSAS-C/P | Change from baseline at 10 weeks
  Is a self-reported scale to measure functional impairment attributed to an identified problem. is a five-item self-report scale measuring functional impairment on a nine-point scale. Higher rating indicating more impairment.
Change of psychiatric symptoms measured with Revised Children's Anxiety and Depression Scale /R-CADS | Change from baseline at 10 weeks
  47-item questionnaires that measure the reported frequency of various symptoms of anxiety and low mood. They produce a total anxiety and low mood score and separate scores for each of the follow sub-scales: separation anxiety; social phobia; generalized anxiety; panic; obsessive compulsive; total anxiety; and, low mood. Each answer being scored on a 4 points Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Blomdahl, PhD, Principal Investigator — Region Vastra Gotaland, Sweden
Locations (1):
- Södra Älvsborgs Hospital, Borås, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No